CLINICAL TRIAL: NCT01357096
Title: Development and Efficacy Evaluation of Integrated Chronic Care and Health Promotion Model for Patients With Coronary Artery Disease in Taiwan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sheng-Hsiung Sheu, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 990179
Record Dates: First submitted 2011-05-18; First posted 2011-05-20 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2010-07

CONDITIONS: Acute Myocardial Infarction; Stable Angina
Keywords: intervention; CABG or PTCA
MeSH Terms: conditions — Angina, Stable

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Comparison group (No Intervention)
  Interventions: Other: Traditional group
- Integrated health care team (Experimental)
  Interventions: Behavioral: Integrated health care team

INTERVENTIONS:
Behavioral: Integrated health care team — CAD education fryers, drugs counseling, diet intervention, individualized exercise program, body weight control, smoking cessation program, and distant CAD care monitoring
  Arms: Integrated health care team
Other: Traditional group — CAD education fryers
  Arms: Comparison group

SUMMARY:
The hypothesis of this project is to examine whether the integrated health care program as the intervention group can reduce the recurrence and mortality of coronary artery-related diseases than the traditional one as the comparison group.

ELIGIBILITY:
Inclusion Criteria:

* patients who suffered from acute myocardial infarction or stable angina with intervention (CABG or PTCA)

Exclusion Criteria:

1. Age > 85 yrs old.
2. Worse short-term prognosis (e.g.cancer, congestive heart failure NYHA IV)
3. Any systemic disease which will limit the exercise program (e.g. bed-ridden stroke)
4. Unable to participate in the trial due to any logic reasons

Max Age: 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
Death, non-fatal MI, non-fatal stroke, recurrent angina, emergency room (ER) visit due to any CV-related diseases or readmission due to any CV-related diseases confirmed by the physicians. | one year

SECONDARY OUTCOMES:
BP, lipid, glucose, EBM drugs and self-care efficacy | one year
  1. Blood pressure < 140/90 mmHg (< 130/80 mmHg in the diabetics and patients with chronic kidney disease)
  2. Hypercholesterolemia：LDL < 100 mg/dl
  3. Diabetic：HbA1c < 7%
  4. Smoking cessation rate
  5. Adherence rate of EBM medication including anti-platelet agent, beta-blocker, RAS blocker and lipid-lowering agent.
  6. Efficacy of self care

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Hospital, Kaohsiung, Taiwan, Taiwan